CLINICAL TRIAL: NCT02129452
Title: Research of Olfactory Neuroepithelial Tissue as a Potential Biomarker of Alzheimer Disease
Brief Title: Olfactory Neuroepithelial Tissue of Alzheimer Disease
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kon Chu, MD, PhD, professor, Seoul National University Hospital
Other Study IDs: 1301056458
Record Dates: First submitted 2014-04-28; First posted 2014-05-02 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Dementia; Neurodegenerative Diseases; Tauopathies; Amyloid beta Peptides; Amyloid Plaque; MicroRNAs; Early Diagnosis
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurodegenerative Diseases; Tauopathies; Plaque, Amyloid; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue including olfactory neuroepithelium from nasal cavity
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- CDR (Clinical dementia rating) 0: 10 participants complaining subjective memory problem and acquiring CDR 0
- CDR 0.5: 10 participants complaining subjective memory problem and acquiring CDR 0.5
- CDR 1: 10 participants with mild cognitive impairment and acquiring CDR 1
- CDR 2: 10 participants with moderate to severe cognitive impairment and acquiring CDR 2

SUMMARY:
The purpose of this study is to evaluate the olfactory neuroepithelium as a biomarker of Alzheimer disease. The early diagnosis of Alzheimer disease is of importance for obtaining better response to treatment, but recently reported biomarkers have some limitations. Olfactory neuroepithelium tissue which is accessible through office-based biopsy without difficulty is known to reflect brain pathology that confirms the diagnosis of Alzheimer disease. This study will help in the early detection and treatment of Alzheimer disease.

DETAILED DESCRIPTION:
Alzheimer disease is the most common form of dementia characterized by insidious onset and slow progression. Pathological changes in the brain of Alzheimer disease (AD) precede clinical symptoms many years, and early treatment provide better outcome. Consequently, detection of AD in early stages is needed. Biologic markers including beta-amyloid and tau protein have been studied for early diagnosis of AD. Recently remarkable biomarkers have drawn attention including CSF proteins and PIB (Amyloid-binding carbon 11-labeled Pittsburgh compound B) PET findings, but they pertain to supportive markers since they reflect brain pathology indirectly.

Postmortem studies of AD patients revealed that beta-amyloid and tau proteins are found in olfactory neuroepithelium and correlate with brain pathological changes. Olfactory neuroepithelium tissue can be obtained through office-based biopsy safely and easily by nasal endoscopy. Especially, early pathological changes of AD can be found in entorhinal cortex and piriform cortex adjacent to olfactory neuroepithelium, this study would be valuable for early detection of AD.

MicroRNAs are small, single-stranded RNA comprising about 20 nucleotides and involved in cell differentiation, growth and death. Recently the investigators reported that microRNA 206 have important role in pathomechanism of AD, thus can be new biomarker and disease-modifying therapeutic target of AD.

Study participants are enrolled from primary care clinic at department of Neurology, Seoul National University Hospital. Patients' clinical presentation, MMSE (Mini mental status exam), CDR (Clinical Dementia Rating) and ADAS-COG-K (Alzheimer Disease Assessment Scale Cognitive Subscale) are collected from routinely executed exams in the clinic. Participants are categorized into four groups according to CDR, and each group enrolls 10 patients respectively. The number of 10 patients per each group was calculated based on previous studies, costs, time and ethical perspectives.

Method for olfactory neuroepithelium biopsy was adopted from Lovell et al. (Arch Otolaryngol. 1982). Concentrations of beta-amyloid and tau proteins are analyzed from ELISA, and microRNA 206 from RT-PCR, northern blot and microarray. These data will be evaluated with clinical features and exam results of participants using general statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* "Probable" Alzheimer disease categorized according to NINCDS-ADRDA criteria
* Written or signed informed consent obtained voluntarily from the subject, or legally acceptable representative(s) in the case of "Vulnerable subjects" with CDR more than 1

Exclusion Criteria:

* Those who are not eligible for nasal cavity biopsy due to behavioral or movement disorder
* Those who are in a hypercoagulable state or who take anticoagulant drugs
* Those who have chronic or active allergic rhinitis which interfere accurate pathological evaluation
* Those who are not suitable for the study to the judgments of researchers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pathological evidence of Alzheimer disease in the olfactory neuroepithelium | Baseline at the time of enrollment. Data will be evaluated in a month.
  beta-amyloid protein, tau protein and micro-RNA 206 concentration according to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Kon Chu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Lee ST, Chu K, Jung KH, Kim JH, Huh JY, Yoon H, Park DK, Lim JY, Kim JM, Jeon D, Ryu H, Lee SK, Kim M, Roh JK. miR-206 regulates brain-derived neurotrophic factor in Alzheimer disease model. Ann Neurol. 2012 Aug;72(2):269-77. doi: 10.1002/ana.23588. PMID 22926857
- [Background] Braak H, Braak E. Neuropathological stageing of Alzheimer-related changes. Acta Neuropathol. 1991;82(4):239-59. doi: 10.1007/BF00308809. PMID 1759558
- [Background] Arnold SE, Lee EB, Moberg PJ, Stutzbach L, Kazi H, Han LY, Lee VM, Trojanowski JQ. Olfactory epithelium amyloid-beta and paired helical filament-tau pathology in Alzheimer disease. Ann Neurol. 2010 Apr;67(4):462-9. doi: 10.1002/ana.21910. PMID 20437581
- [Background] Dubois B, Feldman HH, Jacova C, Dekosky ST, Barberger-Gateau P, Cummings J, Delacourte A, Galasko D, Gauthier S, Jicha G, Meguro K, O'brien J, Pasquier F, Robert P, Rossor M, Salloway S, Stern Y, Visser PJ, Scheltens P. Research criteria for the diagnosis of Alzheimer's disease: revising the NINCDS-ADRDA criteria. Lancet Neurol. 2007 Aug;6(8):734-46. doi: 10.1016/S1474-4422(07)70178-3. PMID 17616482
- [Background] Attems J, Jellinger KA. Olfactory tau pathology in Alzheimer disease and mild cognitive impairment. Clin Neuropathol. 2006 Nov-Dec;25(6):265-71. PMID 17140156
- [Background] Lovell MA, Jafek BW, Moran DT, Rowley JC 3rd. Biopsy of human olfactory mucosa. An instrument and a technique. Arch Otolaryngol. 1982 Apr;108(4):247-9. doi: 10.1001/archotol.1982.00790520047013. PMID 7073597
- [Background] Wrobel BB, Mazza JM, Evgrafov OV, Knowles JA. Assessing the efficacy of endoscopic office olfactory biopsy sites to produce neural progenitor cell cultures for the study of neuropsychiatric disorders. Int Forum Allergy Rhinol. 2013 Feb;3(2):133-8. doi: 10.1002/alr.21080. Epub 2012 Nov 28. PMID 23192985